CLINICAL TRIAL: NCT00253799
Title: Prospective, Single Arm, Pilot Study Evaluating the Safety and Efficacy of Hyaluronan (Hylan GF-20) in Patients With Painful Shoulder Osteoarthritis
Brief Title: A Safety Study of Hylan GF-20 to Treat Shoulder Osteoarthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northwestern Ophthalmic Institute S.C. (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0133-003
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2007-06-25 (Estimated); Status verified 2007-06

CONDITIONS: Painful Shoulder Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Hylan GF-20

SUMMARY:
The objective is to assess the safety and efficacy (over the course of 26 weeks) of 2 intra-articular (IA) Hylan GF-20 (Synvisc) injections in addition to customary care in patients with painful glenohumeral osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* • Be will and able to provide written informed consent prior to any study-related procedures being performed and able to understand and comply with the requirements of this study.

  * Agree to receive fluoroscopically guided injections.
  * Be men or women aged 35 years or older.
  * If female and of childbearing age, must have a negative pregnancy test and have taken oral contraceptives for at least one month prior to treatment and continue for the duration of the study (up to and including the final study visit) or agree to use 2 forms of contraception; otherwise females must be surgically sterile or postmenopausal for at least one year.
  * Have painful, non-inflammatory unilateral osteoarthritis of the shoulder. OA in the contralateral shoulder is permissible provided that the OA symptoms are greater in the study joint. The presence of soft tissue pathology (e.g., rotator cuff tear) is permitted, and will be evaluated by an MRI (taken within 6 months of study entry).
  * Report an initial visual analogue pain score (VAS) of ≥ 30 and ≤ 80.
  * Have radiographic confirmation of osteoarthritis of the shoulder prior to baseline (modified Kellgren and Lawrence Numerical Grading System Grades II - IV) on radiographs performed within 12 weeks of screening
  * Have pain from shoulder OA requiring frequent (> 3 days/week) use of analgesics or NSAIDs for at least 8 weeks prior to screening.

Exclusion Criteria:

* • Pregnant, lactating, or unwilling to use adequate contraception.

  * Prior viscosupplementation in target shoulder joint within 1 year of study entry.
  * Known sensitivity to avian protein or any components of hyaluronan based infection devices, steroids, lidocaine.
  * Known Sensitivity to contrast agent.
  * Used systemic steroids or have had an intra-articular steroid injection in the target shoulder within the last 3 months.
  * Rapidly progressive disease.
  * Acute disease or trauma leading to osteoarthritis of the joint within 2 years of study entry.
  * Presence of a primary inflammatory arthropathy (e.g., rheumatoid, psoriatic, or gouty arthritis).
  * Active skin or soft tissue infection in the area of the injection site.
  * Cervical spin disorders (e.g., radiculopathy) that have been symptomatic and required active treatment within the past 3 months.
  * Any active musculoskeletal condition that would impede measurement of the efficacy of the target shoulder joint (such as fibromyalgia).
  * Any major surgery, arthroplasty or arthroscopy in the target shoulder within 26 weeks of screening or planned surgery within the duration of the study.
  * Septic arthritis in any joints within 3 months prior to screening; any history of septic arthritis in the target shoulder.
  * Any significant chronic skin disorders that could interfere with the evaluation of the injection site.
  * Uncontrolled diabetes mellitus, diabetic neuropathy or infectious complications.
  * Active malignancy receiving treatment.
  * Taking warfarin or parental anticoagulant therapy.
  * Active asthma that may require periodic treatment with steroids during the study period.
  * Use of investigational drug, device, or biologic within 12 weeks of screening
  * Patients with ongoing litigation or workman's compensation claim.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2005-12

PRIMARY OUTCOMES:
-Change from baseline to week 26 evaluation of patient's assessment of pain (VAS rest, motion, night)
-Change from Baseline to follow-up in overall pain and function (WOMAC shoulder rating questionnaire)

SECONDARY OUTCOMES:
-Absolute change in passive range of motion, in flexion, abduction, internal and external rotation
-Requirements for rescue medication use for pain of the shoulder at each scheduled visit

CONTACTS AND LOCATIONS:
Overall Officials: Victoria A Brander, MD, Principal Investigator — Northwestern Ophthalmic Institute S.C.